CLINICAL TRIAL: NCT00714974
Title: A Prospective, Randomized, Blinded Study of BIS Analysis in ICU Patients Requiring Neuromuscular Blocking Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Edward J. Kimball MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UU7643
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: ICU Patients
Keywords: Neuromuscular blocking agents; Bispectral analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Standard of care
- 2 (Experimental): Sedation based on BIS value, oer treating physician discretion.
  Interventions: Device: BIS

INTERVENTIONS:
Device: BIS — Sedation dosing based on BIS value, oer treating physician discretion.
  Arms: 2

SUMMARY:
This is a prospective, randomized, blinded study in which patients will be enrolled into either treated(BIS group) or untreated (non-BIS) group employing bispectral analysis to measure the level of sedation/analgesia in patients receiving neuromuscular blocking agents.

To collect pertinent data on critically ill patients while they are receiving NMBA's. In particular to correlate sedation/analgesic medication needs between a group whose medication use is determined by the values obtained by bispectral analysis to a group who will have medications delivered by the standard of care presently used in the intensive care unit in which they are being treated.

To document that patients who are monitored with bispectral analysis are able to achieve an appropriate level of consciousness in a shorter time and require less manipulation and amounts of sedative or analgesic medications than those who are not monitored.

DETAILED DESCRIPTION:
This is a prospective, randomized and blinded study being done in order to help evaluate the level of consciousness with bispectral analysis (BIS) in ICU patients who are pharmacologically paralyzed with NMBAs (neuromuscular blockade agents) and to assess such things as the amount of time required to achieve the appropriate level of sedation/analgesia. Data will be collected and evaluated via this FDA approved equipment. The intent of this project is to evaluate this technology in those who are requiring "anesthesia" like states (use of NMBAs) for prolonged periods in the critically ill patient population.

ELIGIBILITY:
Inclusion Criteria:

* Consented ICU patient, receiving neuromuscular blocking agents.

Exclusion Criteria:

* Unable to be consented

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2000-02; Primary Completion 2003-02 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Amount of sedation required. | During period of neuromuscular blockade use in ICU

SECONDARY OUTCOMES:
Time requiring neuromuscular blockade and mechanical ventilation. | Time in ICU